CLINICAL TRIAL: NCT06969781
Title: Exploratory Clinical Study on Microwave Ablation With or Without Furmonertinib for Early-Stage Non-Small Cell Lung Cancer
Brief Title: MWA With or Without Furmonertinib for Early-Stage Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shanghai Allist Pharmaceuticals Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Jiayuan Sun, Chief Physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS25074
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TKI-MWA-TKI (Experimental): In the Furmonertinib induction followed by microwave ablation (TKI-MWA-TKI) group, patients first undergo a 3-month induction therapy with the targeted agent. After completion of induction therapy, CT re-examination is performed to assess changes in the lesion. If no contraindications are present, microwave ablation (MWA) is conducted. Post-procedure, in the absence of significant complications, targeted therapy is resumed and continued for up to 21 months, provided no severe toxicities occur.
  Interventions: Device: MWA; Drug: TKI
- MWA-TKI (Experimental): In the microwave ablation combined with Furmonertinib (MWA-TKI) group, microwave ablation (MWA) is initially performed on the lesion. In the absence of significant postoperative complications, targeted therapy is initiated and continued for up to 24 months, provided no severe toxicities occur.
  Interventions: Device: MWA; Drug: TKI
- MWA (Active Comparator): In the MWA group, only microwave ablation (MWA) is performed on the lesion without administration of Furmonertinib.
  Interventions: Device: MWA

INTERVENTIONS:
Device: MWA — Enrolled participants undergo microwave ablation (MWA) after comprehensive assessment of lesion location, size, and individual condition. CT or other imaging modalities are used to monitor changes in the ablation zone. The puncture needle is appropriately distributed within the lesion based on its morphology, and ablation duration is determined by imaging-confirmed coverage of the lesion. All procedures are performed under general anesthesia. Ablation time, power, and cycles are recorded intraoperatively, with continuous ECG monitoring throughout. Immediate post-procedure chest CT or other imaging is performed to document intraoperative complications (e.g., pneumothorax, bleeding). Participants are routinely observed for 24 hours post-procedure, followed by CT re-examination and documentation of any complications.
Drug: TKI — 1. Study Drug: Furmonertinib (Shanghai Allist Pharmaceuticals Co.,Ltd.);
  2. Administration: Oral, 80 mg once daily. In the MWA-TKI group, targeted therapy is initiated post-MWA if no significant complications occur, continuing for up to 24 months without severe toxicity. In the TKI-MWA-TKI group, a 3-month induction with Furmonertinib is followed by CT re-evaluation; if no contraindications are present, MWA is performed, and targeted therapy resumes post-procedure, continuing for up to 21 months without severe toxicity.
  Arms: MWA-TKI; TKI-MWA-TKI

SUMMARY:
This is a single-center randomized trial that investigates microwave ablation (MWA) combined with EGFR-TKI therapy in 120 early-stage NSCLC patients (T1-T2N0M0, EGFR-mutant) unsuitable for standard treatments. Participants are stratified by tumor characteristics and randomized equally to MWA alone, MWA-TKI concurrent, or TKI induction followed by MWA-TKI, assessing disease-free survival, overall survival, and safety outcomes. The study compares the clinical benefits and optimal sequencing of local ablation with targeted therapy in early-stage EGFR-mutant NSCLC management.

DETAILED DESCRIPTION:
This is a single-center, randomized, controlled, exploratory study enrolling patients with mixed ground-glass or solid lesions on CT, histologically or cytologically confirmed as NSCLC, harboring EGFR mutations, and clinically staged as Ia, Ib, or IIa (size ≤5 cm, T1-T2N0M0). Patients deemed unsuitable for or refusing surgery/radiotherapy after multidisciplinary assessment were included. Eligible participants who provided informed consent were randomized in a 1:1:1 ratio into three groups: microwave ablation alone (MWA), MWA combined with targeted therapy (MWA-TKI), or targeted therapy induction followed by MWA combined with targeted therapy (TKI-MWA-TKI). Randomization was stratified by solid tumor proportion (<50% vs ≥50%), tumor size (8-30 mm vs >30 mm), and EGFR mutation status (Ex19del vs Ex21 L858R). The study aims to enroll 120 participants. The primary endpoints include disease-free survival (DFS), overall survival (OS), and the incidence of adverse events. The study evaluates the efficacy, safety, and clinical benefits of MWA combined with EGFR-TKI therapy in early-stage NSCLC, comparing different treatment sequences.

ELIGIBILITY:
Inclusion Criteria:

* CT findings showing mixed ground-glass or solid lesions, histologically or cytologically confirmed as NSCLC, with clinical stages Ia, Ib, or IIa (size ≤5 cm, T1-T2N0M0) according to the 9th edition of TNM classification.
* EGFR exon 19 deletion or exon 21 L858R mutation.
* Age ≥18 years.
* ECOG PS score of 0-2.
* Expected survival ≥3 months.
* Deemed unsuitable for or refusal of surgery/radiotherapy after multidisciplinary discussion.
* No prior EGFR-TKI targeted therapy.
* Willing to undergo initial ablation therapy, with good compliance to examinations and follow-ups, and able to understand the study and provide informed consent.

Exclusion Criteria:

* Severe liver, kidney, heart, lung, or brain dysfunction or other comorbidities that preclude tolerance to MWA or targeted therapy.
* Chest CT findings indicating percutaneous inaccessibility of the lung lesion for MWA.
* Platelet count <50×10⁹/L, severe bleeding tendency, or uncorrectable coagulation disorders.
* Current or prior (within 3 months) use of anti-tumor drugs or EGFR-TKI therapy.
* Uncontrolled conditions (including but not limited to non-pulmonary malignancies, active infections, symptomatic congestive heart failure, unstable angina, arrhythmias, psychiatric disorders, etc.).
* Pregnant or breastfeeding women, or those planning pregnancy during the study.
* Other conditions deemed by the investigator as unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival (DFS) rate in the MWA-TKI and TKI-MWA-TKI groups | From the time of treatment to the time of disease progression or death, assessed up to 3 year
  The proportion of subjects who remain free from disease recurrence or death from the start of treatment until 3 years post-treatment.

SECONDARY OUTCOMES:
1-year and 2-year disease-free survival (DFS) rates in the MWA-TKI and TKI-MWA-TKI groups | From the time of treatment to the time of disease progression or death, assessed up to 1 year or 2 year
  The proportion of subjects who remain free from disease recurrence or death from the start of treatment until 1year post-treatment or 2 years post-treatment.
1-year, 2-year, and 3-year overall survival (OS) rates in the MWA-TKI and TKI-MWA-TKI groups | From the time of treatment to the time of death, assessed up to 1 year, 2 year and 3 year.
  The proportion of subjects who remain alive from the start of treatment until 1 year, 2 years, and 3 years post-treatment.
Overall survival (OS) in the MWA-TKI and TKI-MWA-TKI groups | From the time of treatment to the time of death, assessed up to 5 year.
  The time from the start of treatment to the subject's death or the last follow-up.
1-year, 2-year, and 3-year disease-free survival (DFS) rates in the MWA group. | From the time of treatment to the time of disease progression or death, assessed up to 1 year, 2 year or 3 year.
  The proportion of subjects who remain free from disease recurrence or death from the start of treatment until 1 year, 2 years, and 3 years post-treatment.
1-year, 2-year, and 3-year overall survival (OS) rates in the MWA group | From the time of treatment to the time of death, assessed up to 1 year, 2 year and 3 year.
  The proportion of subjects who remain alive from the start of treatment until 1 year, 2 years, and 3 years post-treatment.
Overall survival (OS) in the MWA group | From the time of treatment to the time of death, assessed up to 5 year.
  The time from the start of treatment to the subject's death or the last follow-up.
The incidence of adverse events (AEs) | 24 months after treatment
  AEs include procedure-related adverse reactions during or after MWA and drug-related adverse reactions caused by targeted therapy.
Exploration of potential predictive biomarkers and synergistic effects of MWA combined with targeted therapy | Disease progression or up to 2 years (whichever occurs first)
  By comparing pre- and post-treatment tumor biopsy specimens, peripheral blood samples, and bronchoalveolar lavage fluid samples, this study investigates changes in local lesions and the systemic microenvironment, including biomarkers, metabolites, and the immune microenvironment, and their relationship with efficacy and prognosis. Additionally, potential regulatory pathways are explored. Furthermore, by comparing the three groups, the study examines whether MWA combined with targeted therapy can produce synergistic effects, whether these effects are related to the timing of targeted therapy, and the underlying regulatory mechanisms of such synergy.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PHD, Principal Investigator — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartlett EC, Rahman S, Ridge CA. Percutaneous image-guided thermal ablation of lung cancer: What is the evidence? Lung Cancer. 2023 Feb;176:14-23. doi: 10.1016/j.lungcan.2022.12.010. Epub 2022 Dec 22. PMID 36571982
- [Background] Herbst RS, Wu YL, John T, Grohe C, Majem M, Wang J, Kato T, Goldman JW, Laktionov K, Kim SW, Yu CJ, Vu HV, Lu S, Lee KY, Mukhametshina G, Akewanlop C, de Marinis F, Bonanno L, Domine M, Shepherd FA, Urban D, Huang X, Bolanos A, Stachowiak M, Tsuboi M. Adjuvant Osimertinib for Resected EGFR-Mutated Stage IB-IIIA Non-Small-Cell Lung Cancer: Updated Results From the Phase III Randomized ADAURA Trial. J Clin Oncol. 2023 Apr 1;41(10):1830-1840. doi: 10.1200/JCO.22.02186. Epub 2023 Jan 31. PMID 36720083
- [Background] Gu XY, Jiang Z, Fang W. Cryoablation combined with molecular target therapy improves the curative effect in patients with advanced non-small cell lung cancer. J Int Med Res. 2011;39(5):1736-43. doi: 10.1177/147323001103900516. PMID 22117974
- [Background] Ni Y, Bi J, Ye X, Fan W, Yu G, Yang X, Huang G, Li W, Wang J, Han X, Ni X, Wei Z, Han M, Zheng A, Meng M, Xue G, Zhang L, Wan C. Local microwave ablation with continued EGFR tyrosine kinase inhibitor as a treatment strategy in advanced non-small cell lung cancers that developed extra-central nervous system oligoprogressive disease during EGFR tyrosine kinase inhibitor treatment: A pilot study. Medicine (Baltimore). 2016 Jun;95(25):e3998. doi: 10.1097/MD.0000000000003998. PMID 27336903
- [Background] Chan MV, Huo YR, Cao C, Ridley L. Survival outcomes for surgical resection versus CT-guided percutaneous ablation for stage I non-small cell lung cancer (NSCLC): a systematic review and meta-analysis. Eur Radiol. 2021 Jul;31(7):5421-5433. doi: 10.1007/s00330-020-07634-7. Epub 2021 Jan 15. PMID 33449192